CLINICAL TRIAL: NCT04812314
Title: Exercise Effects on Adipose Tissue Structure and Function
Acronym: LG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jeffrey F Horowitz, professor of Movement Science and director of the Substrate Metabolism Laboratory (SML) at the University of Michigan School of Kinesiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00175528
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Metabolic Syndrome; Metabolic Disease; Insulin Resistance; Weight Loss; Weight Gain
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Metabolic Diseases; Insulin Resistance; Weight Loss; Weight Gain | interventions — Exercise; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise (Experimental): This exercise prescription represents a common or "conventional" form of physical activity (e.g., moderate/brisk walking). If assigned to this group, participants will perform 45 minutes of moderate intensity continuous steady-state exercise at 70% maximal heart rate (HRmax) to expend 250 calories 4 days per week.
  Interventions: Behavioral: Exercise
- No exercise (Experimental): Subjects assigned to this group are to remain sedentary (no planned physical exercise) throughout the duration of the study.
  Interventions: Behavioral: No exercise

INTERVENTIONS:
Behavioral: Exercise — Participants will complete a moderate intensity continuous exercise 4 days/week.
  Arms: Exercise
Behavioral: No exercise — Participants will remain sedentary throughout the duration of the study.
  Other Names: Control group
  Arms: No exercise

SUMMARY:
Participants will be randomized into one of two different experimental groups: 1) Exercise group and 2) No exercise (control group). Subject participation in the study will involve a series of metabolic tests before and after participants undergo a 10% weight loss program (with or without exercise training depending on group randomization). After completing this weight loss portion of the study, participants will then be required to adhere to a high calorie diet program to regain half of the weight the participant lost - followed by the same series of metabolic tests.

DETAILED DESCRIPTION:
Exercise is among the first line treatments for obesity and obesity-related diseases, yet it is shocking how little is known about how exercise works to improve health. Expanding the knowledge about novel exercise-induced adaptations in fat tissue of obese individuals and furthering the understanding about mechanisms underlying these adaptations could lead to innovative approaches for preventing and treating insulin resistance and obesity-related diseases.

Overall, the researchers believe that exercise training modifies key processes in subcutaneous fat tissue that may contribute to an increase body fat storage capacity (without increasing fat mass). The research team anticipates that exercise will evoke an even more potent adaptive response when fat tissue is dynamically changing in response to alterations in nutritional status (i.e., weight loss and weight regain).

Participants will be randomized into one of two different experimental groups: 1) Exercise group and 2) No exercise (control group). Subject participation in the study will involve a series of metabolic tests before and after participants undergo a 10% weight loss program (with or without exercise training depending on group randomization). After completing this weight loss portion of the study, participants will then be required to adhere to a high calorie diet program to regain half of the weight the participant lost - followed by the same series of metabolic tests. After the participant completes the study, the study team will help the participant to lose more weight. Total involvement in the study for each participant will likely be about 8-10 months.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-40
* Body Mass Index: 27-45 kg/m2
* No regularly planned exercise/physical activity for at least 6 months
* Women must have regularly occurring menses and must be premenopausal

Exclusion Criteria:

* Evidence/history of cardiovascular or metabolic disease
* Medications known to affect lipid or glucose metabolism, or inflammation
* Weight instability ≥ ± 6 pounds in the last 3 months
* Tobacco or e-cigarette users
* Women must not be pregnant or actively lactating

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Oral Glucose Tolerance Test (OGTT) | 2 hours
  A test in which glucose is given and blood samples taken afterward to determine how quickly it is cleared from the blood will be completed at each clinical visit appointment..
Adipose Tissue Fibrosis | 30 minutes
  measured histologically using Sirus Red Staining, quantified using ImageJ software at each clinical visit appointment.
Muscle Capillarization | 30 minutes
  measured immunohistochemically using an antibody for CD31, quantified using ImageJ software at each clinical visit appointment.
Adipose Capillarization | 30 minutes
  measured immunohistochemically using an antibody for CD31, quantified using ImageJ software at each clinical visit appointment.
Fat Cell Size | 3 minutes
  measured histologically using Hematoxylin and eosin (H & E) staining, quantified using ImageJ software at each clinical visit appointment.

SECONDARY OUTCOMES:
Blood Lipid Profile | 15 minutes
  A panel of blood tests that screens for abnormalities in blood lipids will be measured at each clinical visit appointment.
Blood Pressure | 10 minutes
  The pressure of circulating blood against the walls of blood vessels will be measured at screening and each clinical visit appointment.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Horowitz, PhD, Principal Investigator — University of Michigan, School of Kinesiology
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.